CLINICAL TRIAL: NCT01210625
Title: A Randomized, Double Blind, Controlled, Dose Ranging Trial to Compare Nutrabiotix Fiber to Psyllium Fiber in Patients Experiencing Constipation.
Brief Title: Starch-entrapped Microspheres [Nutrabiotix Fiber] for Gut Health
Acronym: NTX
Status: No longer available | Type: Expanded Access
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: Nutrabiotix
Record Dates: First submitted 2010-09-23; First posted 2010-09-28 (Estimated); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Constipation
Keywords: Constipation
MeSH Terms: conditions — Constipation | interventions — Psyllium

INTERVENTIONS:
Dietary Supplement: Nutrabiotix — Fiber supplement: 9mg or 12mg
Dietary Supplement: Psyllium — 12g total per day (4 capsules containing 1 gram psyllium fiber 3 times a day)

SUMMARY:
The investigators hypothesize that daily oral intake of starch-entrapped alginate microspheres (called Nutrabiotix fiber) is well tolerated, exhibits no or minimal "typical" side effects of fiber (e.g. bloating, loose stool, flatulence), can be used as an ideal vehicle to deliver anti-oxidants/anti-inflammatory natural and synthetic substances/agents; and promote gut health by improving bowel habit, by changing the gut microbiota and increasing production of short chain fatty acids, especially butyrate, in the colon and decreasing production of protein putrification (prebiotic effects).

DETAILED DESCRIPTION:
The long-term objective of our research program is to show that targeted colonic delivery of natural specific fermentable carbohydrates will maintain and promote gut health by changing the gut microbiota [prebiotic effect], by increasing "protective and growth promoting" factors such as butyrate, and enhancing intestinal barrier function. These health-promoting functions may prevent and treat a wide range of disorders associated with an abnormal microbiota (dysbiosis) and/or disrupted gut barrier function. Examples of disorders associated with dysbiosis and disrupted gut barrier (leaky gut) are allergic disorders, inflammatory bowel disease, diverticular disease, colon polyps and cancer, alcoholic liver disease, non-alcoholic steatohepatitis (NASH- the most common liver disease in the USA), and irritable bowel syndrome (IBS, the most common GI illness in the US with a high loss of productivity and a high rate of utilization of health care resources).

Nutrabiotix fiber is a prebiotic and is able to promote gut health through changes in the stool microbiota composition favoring saccharolytic bacteria like Bifidobacteria and diminishing proteolytic bacteria like Clostridia. This change in the intestinal microbiota composition should result in increases in the products of carbohydrate fermentation [SCFA] and decreases in the products of protein breakdown [indoles and phenols] in the stool. Also, the fiber is well tolerated and without side effects and is an effective fiber that increases stool bulk and regulates bowel movement.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, asymptomatic 18 to 65 years subjects with BMI 20-30 and self described unsatisfactory bowel habit

Exclusion Criteria:

1. Abnormalities in CBC (Hgb <12 g/dL, platelet count <100 000, WBC <4000 or >10 000);
2. Abnormal liver function tests (ALT, AST, alkaline phosphatase, or bilirubin >1.5 times normal range);
3. Abnormal renal function tests (BUN or creatinine >1.5 times normal range);
4. Low serum albumin (<3 g/dL);

5) Abnormal TSH level;

(6) High CRP;

(7) Significant GI symptoms (except for constipation or occasional rectal bleeding due to hemorrhoids);

(8) Prior intestinal resection;

(9) Patient history of GI diseases [except for hemorrhoids or occasional (<3 times a week) heartburn];

(10) Antibiotic use within last 12 weeks prior to enrollment;

(11) Lean (BMI <25) or obese (BMI>30) subjects because obesity could be associated with abnormal microbiota;

(12) Significant cardiac or respiratory diseases (defined by requiring daily medication for management of their diseases);

(13) Severe hypertension (defined as uncontrolled hypertension in spite of therapy, or requirement of more than one medication to treat hypertension; well-controlled, mild hypertension may be included);

(14) Insulin-requiring and/or poorly controlled diabetes (well-controlled diabetics with HbA1c <6 may be enrolled);

(15) Significant psychological disorders;

(16) Drug and/or alcohol abuse;

(17) Unwillingness to consent to the study;

(18) Plan to have a major change of the dietary habit during the following 5 months;

(19) Subjects younger than 18 or older than 65. Older subjects are excluded in this initial study because of high co-morbidity in older subjects. Children are excluded for this initial Phase I study where the safety is not established;

(20) Pregnant and lactating women due to lack of information about safety of the product in pregnant and lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Michael Brown, M.D., Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Rasmussen HE, Hamaker B, Rajan KB, Mutlu E, Green SJ, Brown M, Kaur A, Keshavarzian A. Starch-entrapped microsphere fibers improve bowel habit but do not exhibit prebiotic capacity in those with unsatisfactory bowel habits: a phase I, randomized, double-blind, controlled human trial. Nutr Res. 2017 Aug;44:27-37. doi: 10.1016/j.nutres.2017.05.015. Epub 2017 Jun 2. PMID 28821315